CLINICAL TRIAL: NCT03298750
Title: Mechanical Stimulation of the Ovary for Infertility Treatment in Patients With Very Low Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-2289-AK-CTIL
Record Dates: First submitted 2016-06-26; First posted 2017-10-02 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Ovarian Stimulation
Keywords: Mechanical Laboratory Ovarian Stimulation Poor responders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mechanical stimulation (Experimental): Mechanical stimulation of ovarian tissue
  Interventions: Procedure: Resection of ovarian tissue and mechanical stimulation

INTERVENTIONS:
Procedure: Resection of ovarian tissue and mechanical stimulation — he women will undergo a surgical laparoscopy during which one of the two technique will ensue.
  1. One of the ovaries will be scratched ( 2 mm depth) with a knife. Simultaneously, a piece of the ovary will be preserved for further histologic analysis and research in the laboratory.
  2. A piece of one ovary will be resected (up to one third of the ovary's volume, without harming the other ovary.
  The resected ovarian tissue will be transferred immediately to the laboratory where the cortex will be divided from the medulla and sliced to small pieces of 1-2 square millimeters.
  These pieces will be transferred back to the operation room in order for them to be transplanted under the serosa layer of the remaining ovary.
  Any bleeding would be stopped using a stiches or hemostatic mesh (diathermy will not be used).
  Simultaneously, a piece of the ovary will be preserved for further histologic analysis and research in the laboratory.

SUMMARY:
Examine the possibility that mechanical stimulation and ovarian fragmentation in women with premature ovarian failure or low ovarian reserve intended for egg donation may cause early follicular recruitment and increase chances of achieving pregnancy through IVF.

DETAILED DESCRIPTION:
The women will undergo a surgical laparoscopy during which one of the two technique will ensue.

1. One of the ovaries will be scratched ( 2 mm depth) with a knife. Simultaneously, a piece of the ovary will be preserved for further histologic analysis and research in the laboratory.
2. A piece of one ovary will be resected (up to one third of the ovary's volume, without harming the other ovary.

The resected ovarian tissue will be transferred immediately to the laboratory where the cortex will be divided from the medulla and sliced to small pieces of 1-2 square millimeters.

These pieces will be transferred back to the operation room in order for them to be transplanted under the serosa layer of the remaining ovary.

Any bleeding would be stopped using a stiches or hemostatic mesh (diathermy will not be used).

Simultaneously, a piece of the ovary will be preserved for further histologic analysis and research in the laboratory.

Post operational follow up ( up to two years) including: menstrual cycle surveillance, hormonal profile, AMH level, US of the pelvis and Antral Follicles Count (AFC).

A month after the surgery, an ovarian stimulation will commence following IVF while close monitoring the ovarian response and comparing the pre and post operation response.

Moreover, the treated ovary will be compared to the untreated one: using the US the ovarian volume and antral follicles size and count will be evaluated.

The preserved pieces of ovary will be histologically evaluated for ovarian reserve analysis.

Additionally, these pieces will be used for experiments for the evaluation of various methods for primordial follicles stimulation including mechanical stimulation like the laser or using substances like Akt Stimulators.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, aged 21-40. with premature ovarian failure.
* Healthy women, with poor ovarian reserve, aged 38-45, undergoing IVF Low ovarian response: recruitment of up to three eggs in previous treatments.
* After the failure of at least 4 cycles.
* Two functioning ovaries, follicular and hormonal response of both ovaries in prior therapies.
* Women candidates for egg donation, and seeking further treatment before switching to egg donation.

Exclusion Criteria:

* Women with kidney disease.
* Women with infertility factors other than ovarian failure, such as endometriosis, PCOS, male factor.
* Women with one non-functioning ovary, or that was removed.
* Women with an intrauterine or pelvic pathology.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-10-20 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Menstrual cycle surveillance | 2 years
  Duration of the menstrual period (days)
AMH | 2 years
  Ovarian reserve measurements. AMH levels ng/ml
Estradiol | 2 years
  Estradiol levels at day of HCG in Pmol/L
Antral follicular count | 2 years
  measurement of. any antral follicles at day 3-5 with ultrasound
IVF outcomes | 2 years
  Number of oocytes at OPU
FSH levels | 2 years
  FSH levels at. day 2-3 of menstruation IU/L
IVF outcomes fertilization rates | 2 years
  fertilization rate. - number of fertilized oocytes relatively to total number of oocytes
IVF outcomes | 2 years
  pregnancy rates

CONTACTS AND LOCATIONS:
Overall Officials: Alon Kedem, MD, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No